CLINICAL TRIAL: NCT02927795
Title: Assessment of Physical Functioning and Handling of Spiolto® Respimat® in Patients With Chronic Obstructive Pulmonary Disease (COPD) Requiring Long-acting Dual Bronchodilation in Routine Clinical Practice
Brief Title: OTIVACTO Spain Non Interventional Study
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1237.58
Record Dates: First submitted 2016-10-06; First posted 2016-10-07 (Estimated); Results first posted 2019-09-30 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Spiolto Respimat: QOL measurement of COPD patients taking Spiolto Respimat

SUMMARY:
This is a self-controlled study design enrolling consented COPD patients who will be treated with Spiolto® Respimat® according to the approved SmPC. Patients will be enrolled consecutively and will be followed over an observational period of approx. 6 weeks.

DETAILED DESCRIPTION:
Purpose:

Study Design:

ELIGIBILITY:
Inclusion criteria:

1. Written informed consent prior to participation
2. Female and male patients = or > 40 years of age
3. Patients diagnosed with Chronic Obstructive Pulmonary Disease (COPD) and requiring long-acting dual bronchodilation (Long-acting muscarinic antagonist (LAMA) + Long-acting beta2 agonist (LABA)) treatment according to approved Spiolto® Respimat® Summary of Product Characteristics (SmPC) and COPD Global Initiative for Chronic Obstructive Lung Disease (GOLD) guideline recommendation

Exclusion criteria:

1. Patients with contraindications according to Spiolto® Respimat® SmPC
2. Patients who have been treated with a LABA/LAMA combination (free and fixed dose) in the previous 6 months
3. Patients continuing Long-acting beta2 agonist and inhalative corticosteroids (LABA-iCS) treatment should not be additionally treated with Spiolto® Respimat® in order to avoid a double dosing of long-acting beta2 agonists
4. Patients for whom further follow-up is not possible at the enrolling site during the planned study period of approx. 6 weeks
5. Pregnancy and lactation
6. Patients currently listed for lung transplantation
7. Current participation in any clinical trial or any other non-interventional study of a drug or device

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients
Sampling Method: Probability Sample
Enrollment: 257 (Actual)
Dates: Start 2017-04-26 (Actual); Primary Completion 2018-09-18 (Actual); Study Completion 2018-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim; Mireia Canals, +34607550925, Study Chair — mireia.canals@boehringer-ingelheim.com
Locations (79):
- Spain (79):
  - Centro de Salud Águilas Sur, Aguilas (Murcia)
  - Consultorio Médico de Albelda, Albelda (Huesca)
  - Centro de Salud Alcantarilla-Sangonera, Alcantarilla (Murcia)
  - Centro de Salud Alquerías Raal, Alquerías (Murcia)
  - Centro de Salud Aranda Norte, Aranda de Duero (Burgos)
  - Centro de Salud Ávila Estación, Ávila
  - Centro de Salud Ávila Rural, Ávila
  - Centro de Salud Ávila Sureste, Ávila
  - Centro de Salud Ávila Suroeste, Ávila
  - Centro de Salud La Paz-Cruces, Barakaldo (Vizcaya)
  - Consulta Privada, Barcelona
  - Centro de Salud de Beniel, Beniel (Murcia)
  - Zorroza Centro de Salud, Bilbao (Vizcaya)
  - Centro de Salud Gazteleku, Bilbao (Vizcaya)
  - Centro Médico IMQ, Bilbao (Vizcaya)
  - Consulta Privada, Bizcaia
  - Centro de Salud Bullas, Bullas (Murcia)
  - Centro de Salud San Agustín, Burgos
  - Centro de Salud Burgos Rural Norte, Burgos
  - Centro de Salud Comuneros, Burgos
  - Centro de Salud Las Torres, Burgos
  - Centre d'Atenció Primària Calella, Calella (Barcelona)
  - Centro de Salud Cartagena Este, Cartagena (Murcia)
  - Centro de Salud Cartagena Oeste, Cartagena (Murcia)
  - Centro de Salud del Barrio de Peral, Cartagena (Murcia)
  - Centre d'Atenció Primària Centelles, Centelles (Barcelona)
  - Centro de Salud de Torrekua, Eibar (Guipúzcoa)
  - Centro de Salud Elgoibar, Elgoibar (Guipuzkoa)
  - Centro de Salud Fuente Álamo, Fuente Álamo (Murcia)
  - C.S. Guardo, Guardo (Palencia)
  - Centro de Salud Sodupe, Güeñes (Vizcaya)
  - Centro de Salud La Unión, La Unión (Murcia)
  - Centro de Salud de Librilla, Librilla (Murcia)
  - Centre d'Atenció Primària Lloret de Mar, Lloret de Mar (Girona)
  - Centro de Salud Joaquín Elizalde, Logroño
  - Centro de Salud Lorca Sur San José, Lorca (Murcia)
  - Centro de Salud San Andrés, Madrid
  - Centre Mèdic Bages, Manresa
  - CS Medina del Campo, Medina del Campo
  - Centro de Salud Medina del Campo Urbano, Medina Del Campo (Valladolid)
  - Centro de Salud Miranda Oeste, Miranda de Ebro (Burgos)
  - Centro de Salud Mula (Consultorio Albudeite), Mula (Murcia)
  - Consultorio Casillas, Murcia
  - Centro de Salud Murcia Sur, Murcia
  - Centro de Salud Murcia-Infante Juan Manuel, Murcia
  - Centro de Salud Espinardo, Murcia
  - Consultorio de Cobatillas, Murcia
  - Centro de Salud Nájera, Nájera (La Rioja)
  - Centro de Salud Oion, Oion (Álava)
  - Consultorio Médico Palazuelos, Palazuelos de Eresma (Segovia)
  - Centro de Salud Pintor Oliva, Palencia
  - Centro Salud Peñaranda de Bracamonte, Peñaranda de Bracamonte (Salamanca)
  - Centro de Salud Castaños, Portugalete (Vizcaya)
  - Pozo Estrecho Centro de Salud, Pozo Estrecho (Murcia)
  - Centro de Salud Quintanar de la Sierra, Quintanar de La Sierra (Burgos)
  - Centro de Salud Universidad Centro de Salamanca, Salamanca
  - Centro de Salud Garrido Sur, Salamanca
  - San Bernado Oeste_Centro de Salud Miguel Armijo, Salamanca
  - Centro de Salud Salvatierra, Salvatierra (Álava)
  - Centro de Salud de Amara Centro, San Sebastián (Guipúzcoa)
  - Centro de Saud Amara-Berri 20010, San Sebastián (Guipúzcoa)
  - Residencia Geriátrica Aldakonea, San Sebastián (Guipúzcoa)
  - Centro de Salud Ambulatorio Gros, San Sebastián (Guipúzcoa)
  - Centro de Salud Santomera, Santomera (Murcia)
  - Centro de Salud Segovia I, Segovia
  - Clínica Médica Goya, Segovia
  - Centro de Salud Segovia II_ La Albuera, Segovia
  - Centro de Salud Markonzaga, Sestao (Vizcaya)
  - Centro de Salud Torre Pacheco, Torre Pacheco (Murcia)
  - Centro de Salud Tudela de Duero, Tudela de Duero (Valladolid)
  - Circunvalación Centro de Salud, Valladolid
  - Centro de Salud Canterac, Valladolid
  - Centro de Salud Casco Viejo, Vitoria (Álava)
  - Centro Médico Medicentro, Vitoria (Álava)
  - C.S. Aranbizkarra I, Vitoria (Álava)
  - Policlínica San José, Vitoria (Álava)
  - Centro de Salud Yecla Oeste, Yecla (Murcia)
  - Centro de Salud Santa Elena, Zamora
  - Centro de Salud Puerta Nueva, Zamora

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Open-label observational study, including Chronic Obstructive Pulmonary Disease (COPD) patients in Spain receiving treatment with Spiolto® Respimat® for approximately 6 weeks, which is the average time between two medical consultations. Questionnaire (quest.).
  10-point increase of Physical functioning questionnaire (PF10 )
Pre-assignment Details: All participants were screened for eligibility to participate in the study. Participants attended primary care centres which would then ensure that all participants met all inclusion/exclusion criteria. Participants were not to be entered if any one of the specific entry criteria were not met.
Groups:
- Spiolto® Respimat®: Chronic Obstructive Pulmonary Disease (COPD) patients were administered a combination of tiotropium and olodaterol in a fixed dose combination through a single Respimat® inhalation device according to approved Summary of Product Characteristics (SPC) and the Global Initiative for Chronic Obstructive Lung Disease (GOLD) guidelines
Period: Overall Study
Arm/Group | Spiolto® Respimat®
Started | 257
Treated | 253
Completed | 234
Not Completed | 23
Not completed — Non-evaluable PF10 quest. at visit 2 | 19
Not completed — Not Treated | 4

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): All screened patients with at least one documented administration of Spiolto® Respimat®.
Arm/Group | Spiolto® Respimat®
Number analyzed (Participants) | 253
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.41 (10.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68
  Male | 185
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Therapeutic Success at Week 6 Approximately (Approx.) (Visit 2)
Description: Therapeutic success defined as at least 10-point increase of Physical functioning questionnaire (PF-10 ) score after approximately 6 weeks of Spiolto® Respimat® treatment. The PF-10 used for assessing the primary outcome "physical functioning" is a subdomain of the validated Short Form 36 (SF-36 ) and consists of 10 questions evaluating the extent of experienced restrictions while conducting usual activities. Each question of the PF-10 can be answered with "yes, limited a lot", "yes, limited a little" or "no, not limited at all", with a score of 1, 2 or 3. The sum of the scores of the 10 questions results in a value between 10 (a patient answering all questions with "yes, limited a lot") and 30 (a patient answering all questions with "no, not limited at all"). The final sum of the individual scores was standardized to a range of 0 to 100 using the following formula: [(sum of scale items - 10) * 100] / 20.
  Higher scores indicate better physical functioning.
Time Frame: After approximately 6 weeks (visit 2)
Population: Full Analysis Set (FAS): All screened patients with at least one documented administration of Spiolto® Respimat® and available PF-10 score at visit 1 and visit 2.
Measure: Number (95% Confidence Interval); unit: Percentage of Patients (%)
Arm/Group | Spiolto® Respimat®
Number analyzed (Participants) | 234
Percentage of Patients (%) | 66.2 [60.2 to 72.3]

2. Secondary Outcome: The Mean Change in the PF-10 Score From Visit 1 (Baseline) to Visit 2
Description: The change in Physical functioning questionnaire (PF-10 ) score was determined by taking into account the individual change of each patient between Baseline (Visit 1) and Week 6 (approx.) (Visit 2) and then the mean for change from baseline values across all patients was calculated.
  The PF-10 consists of 10 questions evaluating the extent of experienced restrictions while conducting usual activities. Each question of the PF-10 can be answered with "yes, limited a lot", "yes, limited a little" or "no, not limited at all", with a score of 1, 2 or 3. The sum of the scores of the 10 questions results in a value between 10 (a patient answering all questions with "yes, limited a lot") and 30 (a patient answering all questions with "no, not limited at all"). The final sum of the individual scores was standardized to a range of 0 to 100 using the following formula: [(sum of scale items - 10) * 100] / 20.
  Higher scores indicate better physical functioning.
Time Frame: Baseline (visit 1) and after approx. week 6 (visit 2)
Population: FAS
Measure: Mean (Standard Deviation); unit: Unit on scale
Arm/Group | Spiolto® Respimat®
Number analyzed (Participants) | 234
Unit on scale | 16.04 (18.18)

3. Secondary Outcome: Patients General Condition Evaluated by the Physician (PGE Score) at Visit 1 and Visit 2
Description: The patient's general condition was evaluated by means of Physician's Global Evaluation (PGE) score. The PGE score is documented on a scale from 1 (poor) to 8 (excellent) at both visits. 1-2: poor; 3-4: satisfactory; 5-6: good; 7-8: excellent
Time Frame: Baseline (visit 1) and after approx.week 6 (visit 2)
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Spiolto® Respimat®
Number analyzed (Participants) | 234
Participants
  Baseline (Visit 1) : PGE score 1 | 2
  Baseline (Visit 1) : PGE score 2 | 48
  Baseline (Visit 1) : PGE score 3 | 57
  Baseline (Visit 1) : PGE score 4 | 49
  Baseline (Visit 1) : PGE score 5 | 35
  Baseline (Visit 1) : PGE score 6 | 31
  Baseline (Visit 1) : PGE score 7 | 7
  Baseline (Visit 1) : PGE score 8 | 5
  Week 6 (approx.) (Visit 2): Score 1 | 1
  Week 6 (approx.) (Visit 2): Score 2 | 5
  Week 6 (approx.) (Visit 2): Score 3 | 14
  Week 6 (approx.) (Visit 2): Score 4 | 42
  Week 6 (approx.) (Visit 2): Score 5 | 46
  Week 6 (approx.) (Visit 2): Score 6 | 83
  Week 6 (approx.) (Visit 2): Score 7 | 36
  Week 6 (approx.) (Visit 2): Score 8 | 7

4. Secondary Outcome: Patient Overall Satisfaction With Spiolto® Respimat® at Visit 2
Description: A patient satisfaction questionnaire on how overall satisfied they were with the Spiolto® Respimat® treatment was also completed during visit 2, using a 7-point ordinal scale, from 1 (very unsatisfied) to 7 (very satisfied).
Time Frame: After approx. 6 weeks (visit 2) of treatment initiation
Population: FAS who completed the questionnaire.14 patients with missing data were excluded from the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Spiolto® Respimat®
Number analyzed (Participants) | 220
Participants
  Very unsatisfied | 0
  Unsatisfied | 2
  Rather unsatisfied | 6
  Neither satisfied, nor unsatisfied | 15
  Rather satisfied | 27
  Satisfied | 127
  Very satisfied | 43

5. Secondary Outcome: Patient Satisfaction With Inhaling From the Respimat® Device
Description: A patient satisfaction questionnaire on how satisfied they were by inhaling with the Respimat® device was also completed during visit 2, using a 7-point ordinal scale, from 1 (very unsatisfied) to 7 (very satisfied).
Time Frame: After approx. 6 weeks (visit 2) of treatment initiation
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Spiolto® Respimat®
Number analyzed (Participants) | 234
Participants
  Very unsatisfied | 1
  Unsatisfied | 3
  Rather unsatisfied | 2
  Neither satisfied, nor unsatisfied | 16
  Rather satisfied | 25
  Satisfied | 129
  Very satisfied | 58

6. Secondary Outcome: Patient Satisfaction With Handling of the Respimat® Inhalation Device
Description: A patient satisfaction questionnaire on how satisfied they were with handling of the Respimat® inhalation device was also completed during visit 2, using a 7-point ordinal scale, from 1 (very unsatisfied) to 7 (very satisfied).
Time Frame: After approx. 6 weeks (visit 2) of treatment initiation
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Spiolto® Respimat®
Number analyzed (Participants) | 234
Participants
  Very unsatisfied | 0
  Unsatisfied | 2
  Rather unsatisfied | 4
  Neither satisfied, nor unsatisfied | 14
  Rather satisfied | 29
  Satisfied | 132
  Very satisfied | 53

ADVERSE EVENTS:
Time Frame: From first drug administration until end of study, up to approx 6 weeks.
Arm/Group | Spiolto® Respimat®
All-Cause Mortality (participants affected / at risk) | 1/253
Serious Adverse Events (participants affected / at risk) | 1/253
Other Adverse Events (participants affected / at risk) | 0/253
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Spiolto® Respimat® (N=253)
Ischaemic stroke (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
The interpretation of the results is limited by the lower number of patients recruited compared to what was planned. Results may not be representative of the Spanish COPD population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2016-06-13): https://cdn.clinicaltrials.gov/large-docs/95/NCT02927795/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-18): https://cdn.clinicaltrials.gov/large-docs/95/NCT02927795/SAP_001.pdf